CLINICAL TRIAL: NCT03729661
Title: Exploratory Study on Nasal High Flow Therapy for Breath Hold in Radiotherapy.
Brief Title: Exploratory Study on Therapy for Breath Hold in Radiotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht Radiation Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ENTheR
Record Dates: First submitted 2018-10-29; First posted 2018-11-05 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2019-12

CONDITIONS: Lung Cancer; Breast Cancer
MeSH Terms: conditions — Lung Neoplasms; Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Exploratory study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Breath hold (Experimental): Patients who receive a breathhold CT- and treatment
  Interventions: Behavioral: Nasal High Flow Therapy

INTERVENTIONS:
Behavioral: Nasal High Flow Therapy — Use of Nasal High Flow Therapy during CT and treatment

SUMMARY:
Due to breathing and other motions, tumours, such as breast and lung cancer, as well as their surrounding organs (e.g. the heart), move, which poses a challenge for radiotherapy treatment. Reducing or even stopping breathing, e.g. by irradiating during inspiration, is a way to decrease tumour and organ motion resulting in a reliable target coverage with smaller margins. These smaller margins can result in a better sparing of normal tissues. Furthermore, in some patients, during inspiration, the heart may move away from the target volume making it possible to better spare the heart. Finally, during inspiration, the lung volume is larger and the lung density is lower, which can lead to a lower dose to the surrounding normal lung tissue. Reduction of radiation dose to normal tissues leads to less radiation-induced toxicity. This makes treating breast and lung cancer patients in breath hold (BH) conditions an attractive strategy. Standard BH durations in RT treatment are around 20 seconds, which is not enough to perform a complete CBCT. The health status of lung cancer patients is generally worse compared to breast cancer patients, making it more difficult to treat this patient group during breath hold. Nasal High Flow Therapy (NHFT) is a non-invasive system that provides controlled oxygen concentrations and low levels of positive pressure via a nasal interface. NHFT improves oxygenation in diverse patient groups, and is increasingly used as an alternative to mechanical ventilatory support. It has been shown to be a safe device in several clinical situations and patient populations, such as COPD patients, but also in apneic conditions under general anesthesia.

DETAILED DESCRIPTION:
Due to breathing and other motion, tumours, such as breast and lung cancer, as well as their surrounding organs (e.g. the heart), move, which poses a challenge for radiotherapy treatment. Reducing or even stopping breathing, e.g. by irradiating during inspiration, is a way to decrease tumor and organ motion resulting in a reliable target coverage with smaller margins. These smaller margins can result in a better sparing of normal tissues. Furthermore, in some patients, during inspiration, the heart may move away from the target volume making it possible to better spare the heart. Finally, during inspiration, the lung volume is larger and the lung density is lower, which can lead to a lower dose to the surrounding normal lung tissue. Reduction of radiation dose to normal tissues leads to less radiation-induced toxicity. This makes treating breast and lung cancer patients in breath hold (BH) conditions an attractive strategy. A BH has to be stable and long enough for the duration of a planning CT-scan, cone beam CT (CBCT) scan and treatment delivery. Treatment of left-sided breast cancer with radiotherapy in moderate deep inspiration breath hold (mDIBH) is well established. Also, in MAASTRO clinic, left-sided breast cancer patients are treated in mDIBH, but this is done without any support or control of the breath hold. Standard BH durations in RT treatment are around 20 seconds, which is not enough to perform a complete CBCT. The health status of lung cancer patients is generally worse compared to breast cancer patients, making it more difficult to treat this patient group during breath hold. mDIBH in lung cancer patients is therefore not widely used, and not yet performed in MAASTRO clinic. Ventilation techniques that can support patients in holding their breath might make it a feasible approach in patients with a less favourable performance status, and might increase the duration of a breath hold. Nasal High Flow Therapy (NHFT) is a non-invasive system that provides controlled oxygen concentrations and low levels of positive pressure via a nasal interface. NHFT improves oxygenation in diverse patient groups, and is increasingly used as an alternative to mechanical ventilatory support. It has been shown to be a safe device in several clinical situations and patient populations, such as COPD patients, but also in apneic conditions under general anesthesia. It has however never been used in the context of breath hold support, neither has it been used in radiotherapy practice. The investigators hypothesize that supporting BH with nasal high flow therapy (NHFT) will allow robust radiotherapy treatments of moving targets in a broad patient population allowing for BHs that are long enough, stable and reproducible during a whole treatment course.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced lung cancer or oligometastatic patients with "local" stage III, treated with curative or radical intent OR
* Left-sided breast cancer patients treated with radiotherapy with curative intent.
* WHO≤ 2
* ≥ 18 years old
* Able to give informed consent

Exclusion Criteria:

* Patient refusal
* Hypercapnic COPD patient (= arterial carbon dioxide tension PaCO2 > 45 mmHg)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-04-18 (Actual); Primary Completion 2020-01-03 (Actual); Study Completion 2020-01-03 (Actual)

PRIMARY OUTCOMES:
Completing proportion (Tolerability) | 40 days
  The proportion of patients completing the treatment (CT-scan and alle treatment sessions) in breath hold conditions using nasal high flow therapy (Tolerability of the treatment)

SECONDARY OUTCOMES:
Poroportion of patients able to complete breathhold during training | 90 seconds
  Proportion of patients in the population, able to do at least one breath hold of at least 90 seconds during the training session, measured by counting the absolute number of patients.
Investigation of the stability of a breath hold. Breath hold is considered stable if the variations during a breath hold are within 3 mm. | 90 seconds
  Investigation of the stability of a breath hold, the position of the chest during the whole duration of the breath hold, monitored by the surface guidance system, installed in the CT and treatment room. Breath hold is considered stable if the variations during a breath hold are within 3 mm.
Reproduciblity of the breath hold | Overall radiation treatment schedule, varies up to 4 weeks.
  The difference between the baseline chest position (during planning breath hold CT scan) and breath hold during each fraction.
Subjective tolerance as commented by volunteers | Overall radiation treatment schedule, varies up to 4 weeks.
  Comments of volunteers after the test will be recorded as free text.
Subjective tolerance | Overall radiation treatment schedule, varies up to 4 weeks.
  Comments of volunteers after the test will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Stéphanie Peeters, Principal Investigator — Maastro Clinic, The Netherlands; Gloria Vilches, Principal Investigator — Maastro Clinic, The Netherlands
Locations (1):
- Maastricht Radiation Oncology, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: No